CLINICAL TRIAL: NCT02888873
Title: Prospective, Randomized, Controlled, Double Blind Trial of Two Universal Composites in Posterior Teeth
Brief Title: Comparison of Two Universal Composites in Posterior Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zeynep Bilge Kutuk, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014/03-13(KA-14005)
Record Dates: First submitted 2016-08-24; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Dental Caries
Keywords: composite resin; Clinical trial; FDI (World Dental Federation) criteria
MeSH Terms: conditions — Dental Caries | interventions — Charisma composite resin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Charisma (Active Comparator): applied randomly
  Interventions: Other: Charisma
- Charisma classic (Active Comparator): applied randomly
  Interventions: Other: Charisma Classic

INTERVENTIONS:
Other: Charisma — The surfaces were etched using 35% phosphoric acid for 30 s. The etched surfaces were rinsed and dried. Charisma was used in combination Gluma2 Bond etch&rinse adhesive. The composite resin restorations were light-cured (600 milliwatt/cm²). Occlusion was checked with thin articulating papers.
  Restoration surfaces were finished and polished with fine finishing diamond burs, stones and rubber cups.
  Other Names: universal composite
  Arms: Charisma
Other: Charisma Classic — The surfaces were etched using 35% phosphoric acid for 30 s. The etched surfaces were rinsed and dried. Charisma classic was used in combination Gluma2 Bond etch&rinse adhesive. The composite resin restorations were light-cured (600 milliwatt/cm²). Occlusion was checked with thin articulating papers.
  Restoration surfaces were finished and polished with fine finishing diamond burs, stones and rubber cups.
  Other Names: universal composite
  Arms: Charisma classic

SUMMARY:
The aim of this randomized, prospective clinical study was to compare the clinical performance of a universal light-curing, ultra-fine particle hybrid composite with a new version of this product produced by the same manufacturer in Class 1 and Class 2 lesions.

DETAILED DESCRIPTION:
A total of 80 (13 Class 1 and 67 Class 2) lesions in 40 patients (21 females, 19 males) with ages ranging between 18-38 years (23.15±5.15) were either restored with Charisma or Charisma Classic (Heraeus Kulzer) in combination with an etch and rinse adhesive system (Gluma 2 Bond) under rubber dam isolation by two experienced operators according to the manufacturer's instructions. Two independent examiners, who were blinded to the composites used evaluated the restorations according to the FDI (World Dental Federation) criteria. Bite-wing radiographs and intraoral digital photographs were taken before and after treatment and at 6 months. The statistical analyses were carried out with McNemar, Pearson Chi-square and Cochran Q tests (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* a need for at least two but not more than four posterior tooth-colored restorations
* the presence of teeth to be restored in occlusion
* teeth that were symptomless and vital
* a normal periodontal status
* a good likelihood of recall availability.

Exclusion Criteria:

* partly erupted teeth
* absence of adjacent and antagonist teeth
* poor periodontal status
* adverse medical history
* potential behavioral problems.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Observers evaluated the esthetic properties of the restorations using FDI (World Dental Federation) Criteria. | The changes at restorations were obtained from baseline (one week after treatment), 6 month, 1, 2, 3 and 4 year.
  "Surface luster"; "Staining (surface, margins)"; "Color match and translucency"; "Esthetic anatomical form"

SECONDARY OUTCOMES:
Observers evaluated the functional properties of the restorations using FDI (World Dental Federation) Criteria. | The changes at restorations were obtained from baseline (one week after treatment), 6 month, 1, 2, 3 and 4 year.
  "Fracture of material and retention"; "Marginal adaptation"

OTHER OUTCOMES:
Observers evaluated the biological properties of the restorations using FDI (World Dental Federation) Criteria. | The changes at restorations were obtained from baseline (one week after treatment), 6 month, 1, 2, 3 and 4 year.
  "Recurrence of caries, erosion, abfraction"; and "Tooth integrity (enamel cracks, tooth fractures)"

CONTACTS AND LOCATIONS:
Overall Officials: Sevil Gurgan, DDS, PhD, Study Director — Hacettepe University School of Dentistry
Locations (1):
- Hacettepe University School of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Gurgan S, Vural UK, Kutuk ZB, Cakir FY. Comparison of two universal composites in posterior teeth: preliminary report. J Dent Res (Spec Iss 94 B): 308, 2015
- [Derived] Gurgan S, Koc Vural U, Kutuk ZB, Cakir FY. Does a new formula have an input in the clinical success of posterior composite restorations? A chat study. Clin Oral Investig. 2021 Apr;25(4):1715-1727. doi: 10.1007/s00784-020-03472-5. Epub 2020 Aug 3. PMID 32748072